CLINICAL TRIAL: NCT01078610
Title: Long Term Documentation of the Safety and Efficacy as Well as the Effects on Quality of Life and Work Productivity in Patients With Psoriatic Arthritis Under HUMIRA® (Adalimumab) in Routine Clinical Practice
Brief Title: Safety and Effectiveness and Effect on Quality of Life and Work Productivity of Humira in Patients With Psoriatic Arthritis in Clinical Routine
Acronym: ELAN
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped prior to enrollment.
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-023
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-06

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Long-term Observation; Humira; Safety; Effectiveness; Quality of Life; Work Productivity
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriatic arthritis patients
  Interventions: Biological: adalimumab (Humira)

INTERVENTIONS:
Biological: adalimumab (Humira) — 40 mg adalimumab (Humira) every other week.
  Other Names: adalimumab; Humira

SUMMARY:
Safety and effectiveness, quality of life and work productivity of Humira in patients with psoriatic arthritis in clinical routine.

DETAILED DESCRIPTION:
The primary objective of the Non-Interventional Study is to explore the therapeutic success, measured by improvements in the following target variables (with regard to the respective baseline value):

* The number of missed working days
* The self-assessed workability
* The severity of clinical symptoms (number of tender and swollen joints, C-reactive Protein and erythrocyte sedimentation rate respectively; total score Disease Activity Score 28, Psoriasis Area and Severity Index)
* The severity of functional impairment (Health Assessment Questionnaire)
* The health-related quality of life .

All of the patient and disease characteristics which are documented at baseline will be evaluated for their additional impact on the target variables (therapeutic success). Particularly the impact of previous biologic therapies on clinical target variables will be evaluated.

The secondary objective is to document the therapeutic success by the following variables:

* The number of physician visit
* The number and duration of hospitalization
* The number of days of impairment in non-occupational activities
* Pain, exhaustion/fatigue
* The reduction of number and dose of concomitant medication
* Patient's assessment of adalimumab therapy compared to previous therapies.

Target parameters for safety evaluation of adalimumab are:

* The evaluation of safety and tolerability by the documentation and analysis of serious adverse events (SAEs) and adverse events (AEs)
* Evaluation of safety and tolerability for subgroups of patients with common frequent concomitant diseases, especially diabetes type II, cardiovascular, liver, and renal insufficiencies, and related concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Active and progressive psoriatic arthritis in adults with insufficient response to prior basic therapy

Exclusion Criteria:

* Hypersensitivity against the drug or one of the other ingredients
* Active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections)
* Moderate to severe cardiac insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample: patients with psoriatic arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Improvement in: number of missed working days, self-assessed workability, severity of clinical symptoms and functional impairment, health-related quality of life; safety an tolerability: documentation of adverse events and serious adverse events | Months 0, 3, 6, 12, 24, 36, 48, 60

SECONDARY OUTCOMES:
Number and duration of hospitalization; reduction of number and dose of concomitant medication: patient's assessment of adalimumab therapy compared to previous therapies. | Months 0, 3, 6, 12, 24, 36, 48, 60

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Simianer, MD, Study Director — Abbott Germany, Medical Department